CLINICAL TRIAL: NCT00892697
Title: #0810010040: Intrahepatic HCV RNA and Telaprevir Kinetics in Hepatitis C Virus Infection: A Study of Telaprevir in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Subjects With Hepatitis C
Brief Title: Intrahepatic HCV RNA and Telaprevir Kinetics in Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0810010040
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C
Keywords: hepatitis C; FNA; intrahepatic
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm (Experimental): 15 subjects will receive Telaprevir in combination with pegylated interferon alfa-2a and ribavirin
  Interventions: Drug: Telaprevir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Fifteen subjects will receive the same treatment: 12 weeks of telaprevir (750 mg q8h) with Peg-IFN- alfa-2a (Pegasys(R)) (180 mcg SQ qwk) and RBV (1200 mg per day if >75 kg or 1000mg per day if < 75 kg).
Drug: Peginterferon alfa-2a — Fifteen subjects will receive the same treatment: 12 weeks of telaprevir (750 mg q8h) with Peg-IFN- alfa-2a (Pegasys(R)) (180 mcg SQ qwk) and RBV (1200 mg per day if >75 kg or 1000mg per day if < 75 kg).
Drug: Ribavirin — Fifteen subjects will receive the same treatment: 12 weeks of telaprevir (750 mg q8h) with Peg-IFN- alfa-2a (Pegasys(R)) (180 mcg SQ qwk) and RBV (1200 mg per day if >75 kg or 1000mg per day if < 75 kg).

SUMMARY:
The purpose of this study is to determine the decline of virus in the blood and liver in patients treated with telaprevir, pegylated interferon and ribavirin.

Fine Needle Aspiration (FNA) procedure will be used to repeatedly sample the liver to enhance the understanding of how the virus decays in the liver in response to treatment with anti-viral compounds and the measurement of the concentration of the drugs in the liver. FNA is an alternative procedure to core needle biopsy in its ability to repeatedly sample the liver with significantly reduced morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 18-65 years of age, inclusive.
2. Cases will be genotype 1 (confirmed by standard testing). Enrollment of controls will not be restricted by genotype.
3. All patients must show evidence of chronic hepatitis C, confirmed by detectable plasma HCV RNA. Chronic disease status must be confirmed by at least one of the following standard criteria:

   History of a remote risk factor, or Abnormal ALT levels for >6 months prior to screening period (Note: elevated ALT is not an inclusion criteria, if one of the other criteria for "chronic" hepatitis C is met), or Detectable HCV RNA for at least 6 months before the screening period
4. Liver biopsy obtained within 24 months of study enrollment demonstrating absence of cirrhosis (stage 0-3) for cases. Enrollment of controls will not be restricted by stage of fibrosis.
5. Judged to be in good health on the basis of medical history and physical examination (including vital signs and ECG), with any chronic medical conditions under stable medical control.
6. Screening Visit laboratory values must be within the following:

   * Laboratory variable: acceptable range
   * Absolute neutrophil count: 1200/cmm³
   * Platelet count: 90,000/cmm³
   * Hemoglobin: within normal range
   * HbsAg (screening visit only): seronegative
   * HIV1 and 2 Ab (screening visit only): seronegative

   In addition, all other hematology and clinical chemistry must be within normal limits or show no clinically significant abnormalities.
7. Subjects (or their female partners) must be not pregnant, planning to become pregnant within the next 72 weeks, or they must be permanently sterile or otherwise of non childbearing potential. They must also not be breastfeeding. If of child-bearing potential, subjects must agree to use 2 effective methods of contraception from screening through 6 months after the last dose of RBV. Male subjects who have a female partner of childbearing potential must agree to use 2 effective methods of contraception from Screening through 7 months after the last dose of RBV unless vasectomized.
8. Female subjects must have a negative pregnancy test at all visits (screening and predose Day 1) before the first dose of study drugs.
9. Willing to refrain from the concomitant use of any medications, substances or foods.
10. Able to read and understand the Informed Consent Form (ICF) and willing to sign the ICF and abide by the study requirements and restrictions.

Exclusion Criteria:

1. Received more than 4 weeks of any approved or investigational drug or drug regimen for the treatment of hepatitis C.
2. Any medical contraindications to Peg-IFN alpa-2a or RBV therapy, including any of the following:

   1. Abnormal thyroid stimulating hormone (TSH) levels or poorly controlled thyroid function
   2. Evidence of clinically significant cardiac dysfunction;
   3. History of psychiatric disorders determined by the investigator to contraindicate the use of IFN-based therapy;
   4. Antinuclear antibody (ANA) titer 1:320;
   5. History of hemoglobinopathies.
3. Patients coinfected with either human immunodeficiency virus (HIV) or hepatitis B virus (HBV).
4. Decompensated liver disease as indicated by a history of ascites, hepatic encephalopathy, or bleeding esophageal varices.
5. Diagnosed or suspected hepatocellular carcinoma. Alfa-fetoprotein (AFP) during screening must be less than 100 ng/mL.
6. For cases, histologic evidence of hepatic cirrhosis on any liver biopsy

   o Most recent liver biopsy must be within 2 years prior to study screening.
7. Has taken any of the prohibited medications within 28 days of initiation of therapy.
8. A history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include but is not limited to a history of relevant drug or food allergies, history of cardiovascular or central nervous system disease, history or presence of clinically significant illness, or history of mental illness that may affect compliance with study requirements.
9. Alcohol abuse or excessive use (in the opinion of the investigator, as judged by medical history) in the last 12 months.
10. Participation in any investigational drug study within 90 days before drug administration or participation in more than 2 drug studies in the last 12 months (exclusive of the current study).
11. For cases, hypersensitivity to tartrazine (known as yellow dye #5).
12. Men whose female partners are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Talal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University

REFERENCES:
- [Result] Talal AH, Dimova RB, Zhang EZ, Jiang M, Penney MS, Sullivan JC, Botfield MC, Chakilam A, Sawant R, Cervini CM, Zeremski M, Jacobson IM, Kwong AD. Telaprevir-based treatment effects on hepatitis C virus in liver and blood. Hepatology. 2014 Dec;60(6):1826-37. doi: 10.1002/hep.27202. Epub 2014 Jul 31. PMID 24811404
- [Derived] Zeremski M, Dimova RB, Benjamin S, Penney MS, Botfield MC, Talal AH. Intrahepatic and Peripheral CXCL10 Expression in Hepatitis C Virus-Infected Patients Treated With Telaprevir, Pegylated Interferon, and Ribavirin. J Infect Dis. 2015 Jun 1;211(11):1795-9. doi: 10.1093/infdis/jiu807. Epub 2014 Dec 15. PMID 25512630

RESULTS

PARTICIPANT FLOW:
Groups:
- Telaprevir/Peg-IFN/RBV: 15 subjects received Telaprevir in combination with pegylated interferon and ribavirin.
  Telaprevir: Fifteen subjects received the same treatment: 12 weeks of telaprevir (750 mg q8h) with Peg-IFN- alfa-2a (Pegasys(R)) (180 mcg SQ qwk) and RBV (1200 mg per day if >75 kg or 1000mg per day if < 75 kg).
Period: Overall Study
Arm/Group | Telaprevir/Peg-IFN/RBV
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Telaprevir/Peg-IFN/RBV
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [46.5 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Intrahepatic and Plasma HCV Viral Kinetics
Description: Intrahepatic viral kinetics, plasma viral kinetics,
Time Frame: Day-7, Day 1, Day 4,
Measure: Mean (Standard Deviation); unit: log transformed copies/ml
Groups:
- Telaprevir/Peg-IFN/RBV: 15 subjects will receive Telaprevir in combination with pegylated interferon and ribavirin and 5 additional subjects on standard of care.
  Telaprevir: Fifteen subjects will receive the same treatment: 12 weeks of telaprevir (750 mg q8h) with Peg-IFN- alfa-2a (Pegasys(R)) (180 mcg SQ qwk) and RBV (1200 mg per day if >75 kg or 1000mg per day if < 75 kg). Additional 5 subjects be on standard of therapy.
Arm/Group | Telaprevir/Peg-IFN/RBV
Number analyzed (Participants) | 15
log transformed copies/ml
  Plasma HCV RNA predose | 6.5 (0.8)
  Plasma HCV RNA 10 hrs | 4.9 (0.9)
  Plasma HCV RNA day 4 | 3.2 (0.6)
  Liver HCV RNA predose | 4.2 (1.2)
  Liver HCV RNA 10 hrs | 4.0 (1.3)
  Liver HCV RNA day 4 | 3.9 (1.2)

2. Secondary Outcome: Intrahepatic and Peripheral Pharmacokinetic Assessment of Telaprevir
Description: Intrahepatic and plasma telaprevir concentration ratios
Time Frame: Day 1, Day 4, Day 15, Week 8
Measure: Median (Inter-Quartile Range); unit: telaprevir liver to plasma conc ratio
Groups:
- Telaprevir/PEG-IFN/RBV: 15 subjects will receive Telaprevir in combination with pegylated interferon alfa-2a and ribavirin
Arm/Group | Telaprevir/PEG-IFN/RBV
Number analyzed (Participants) | 15
telaprevir liver to plasma conc ratio
  telaprevir liver/plasma conc ratio day 1 | 0.72 [0.4 to 1.01]
  telaprevir liver/plasma conc ratio day 4 | 0.47 [0.33 to 0.78]
  telaprevir liver/plasma conc ratio day 15 | 0.57 [0.34 to 0.76]
  telaprevir liver/plasma conc ratio week 8 | 0.61 [0.42 to 0.84]

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 24 weeks post treatment cessation.
Arm/Group | Telaprevir/PEG-IFN/RBV
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telaprevir/PEG-IFN/RBV (N=15)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telaprevir/PEG-IFN/RBV (N=15)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No